CLINICAL TRIAL: NCT06791733
Title: The Effects of Inter-set Stretching on Muscle Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Luca Di Bartolo, PhD Student, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 150/2023; University of Palermo (Other: University of Palermo)
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AN (Experimental): Participants will perform passive static stretching of antagonist muscles (dorsal muscles) between sets.
  Interventions: Other: Passive static stretching
- AG (Experimental): Participants will perform passive static stretching of agonist muscles (pectoralis muscles) between sets.
  Interventions: Other: Passive static stretching
- CG (No Intervention): Participants will not perform any stretching between sets.

INTERVENTIONS:
Other: Passive static stretching — the intervention consists of passive static stretching of agonist or antagonist muscles between sets
  Arms: AG; AN

SUMMARY:
Static passive muscle stretching, performed weekly, can increase muscle flexibility and range of motion. Typically, static stretching is performed either before starting specific exercises or at the end of a workout. However, the effects of static passive stretching when performed during sets are still not entirely clear in terms of performance. This study aims to evaluate the effects of inter-set stretching on muscle performance

DETAILED DESCRIPTION:
This project aims to evaluate the potential effects of stretching exercises on muscular performance. In particular, we aim to administer passive static stretching between sets of a bench press performance. Within this project we will carry out a crossover design project in which the participants will be tested for two conditions and one control session. The main protocol consists of performing five sets of bench press at 70% of 1-RM. The 1-RM will be calculated before the start of the data collection procedure, through a standardized and validated approach. The experimental sessions will comprise two interventions. The first intervention will be to administer the stretching protocol to the agonist muscles involved in the bench press performance (pectoralis muscles). While the second intervention will be to administer the stretching protocol to the antagonist muscles involved in the bench press performance (dorsal muscles). Within the control session the participants will not perform any stretching between sets. The three arms will be randomized. As outcome variables, the primary outcome will be the comparison of the total volume across each agonist, antagonist, and control session. The secondary outcomes to be assessed are strength, power, velocity, and volume.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged ≥ 18 years.
* At least 6-month experience of resistance training.
* No previous musculoskeletal injuries in the 6 months prior to the study will be recruited

Exclusion Criteria:

* Participants who suffered an injury within the 6 months prior to the study and/or participants with pathological conditions affecting the musculoskeletal system will not be recruited.
* Female participants
* Participants with less than 18 years.
* Participants who match all inclusion criteria but who fail to attend one or more of the agonist/antagonist stretching sessions will be also excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscular performance | From enrollment to the end of a treatment at 2 weeks
  The total volume across each agonist, antagonist, and control session

SECONDARY OUTCOMES:
Strength | From enrollment to the end of a treatment at 2 weeks
  Strength, measured in Newtons, will be evaluated using the 'T-Force' device, which records and collects the main biomechanical parameters, including strength, during the concentric and eccentric phases of movement.
Power | From enrollment to the end of a treatment at 2 weeks
  Power, measured in Watts, will be evaluated using the 'T-Force' device, which records and collects the main biomechanical parameters, including power, during the concentric and eccentric phases of movement.
Velocity | From enrollment to the end of a treatment at 2 weeks
  Velocity, measured in meters per second, will be evaluated using the 'T-Force' device, which records and collects the main biomechanical parameters, including velocity, during the concentric and eccentric phases of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon reasonable request of the corresponding author